CLINICAL TRIAL: NCT00151359
Title: Clinical Trials Stage of 'SoleSensor': A Balance-Enhancing Shoe Insert.
Status: Completed | Type: Observational
Sponsor: Wilfrid Laurier University (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other)
Other Study IDs: PPP-53686
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2005-09-08 (Estimated); Status verified 2005-09

CONDITIONS: Sensation Disorder
MeSH Terms: conditions — Sensation Disorders

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Device: SoleSensor

SUMMARY:
Our research has shown that pressure sensation from the soles of the feet (plantar mechanoreceptors) plays an important role in controlling several key aspects of balancing reactions, particularly during compensatory stepping . As a result, age-related loss of plantar pressure sensation, which is very common, can lead to impaired control of these reactions. However, we have shown that it is possible to compensate for balance impairments resulting from this loss of sensation by using special footwear insoles to facilitate sensation from the perimeter of the sole. To date, we have demonstrated the feasibility of this approach in laboratory studies, and we have obtained a U.S. patent for the design concept. However, it remains to be determined whether the benefits of the footwear persist over the long term, or whether there is a habituation of the effect. Also, we need to determine whether there are any practical problems associated with wearing such footwear, e.g. due to discomfort or irritation of the skin.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 to 75 years

Exclusion Criteria:

* Any neurological or musculoskeletal ailments that affect their balance
* Any drugs that affect balance

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Dates: Start 2002-02

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D Perry, PhD, Principal Investigator — Wilfrid Laurier University; Brian E Maki, PhD, Principal Investigator — Centre for Studies In Aging, Sunnybrook & Women's; Geoff R Fernie, PhD, Principal Investigator — Centre for Studies In Aging, Sunnybrook & Women's
Locations (1):
- WLU Biomechanics Laboratory, Waterloo, Ontario, Canada

REFERENCES:
- [Background] Perry SD, Santos LC, Patla AE. Contribution of vision and cutaneous sensation to the control of centre of mass (COM) during gait termination. Brain Res. 2001 Sep 14;913(1):27-34. doi: 10.1016/s0006-8993(01)02748-2. PMID 11532244